CLINICAL TRIAL: NCT00746993
Title: Structured Contraceptive Counseling--A Randomized Controlled Trial
Brief Title: Randomized Controlled Trial of Structured Contraceptive Counseling in Adult Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Carolyn L. Westhoff, Professor of Obstetrics and Gynecology, Population and Family Health and Epidemiology at the New York-Presbyterian Hospital at the Columbia University Medical Center, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AAAD5101
Record Dates: First submitted 2008-09-02; First posted 2008-09-04 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Contraception
Keywords: Contraception; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Structured contraceptive counseling and routine care.
  Interventions: Other: Structured contraceptive counseling
- 2 (No Intervention): Routine care.

INTERVENTIONS:
Other: Structured contraceptive counseling — Uniform set of visual information about contraception which a counselor will read out loud with each participant and answer questions.
  Other Names: Family Planning Decision Making Tool
  Arms: 1

SUMMARY:
In the United States, highly effective methods of birth control are often not used. Healthcare providers use birth control counseling and patient education as ways to increase the usage of birth control. However, little evidence exists to show that patient education and birth control counseling changes birth control use.

We want to evaluate the effectiveness of using a uniform set of birth control information to provide birth control education to women having an early pregnancy termination. The counselors will allow the clients to both read as well as hear the information. We propose to evaluate whether this counseling will lead to 1) more women choosing highly effective nonpermanent birth control methods and 2) more women continuing to use these methods for a longer time.

Women in the study will complete a questionaire about their health. Half of them will have the structured counseling and half will have the routine counseling currently offered to women as a part of their routine care. We will contact all study participants with a telephone call three months and six months later to have a 10 minute conversation about what birth control they are using.

DETAILED DESCRIPTION:
The proposed study will be a randomized controlled trial to evaluate the primary study hypothesis that structured counseling immediately before a first trimester vacuum aspiration procedure will result in more women choosing a highly effective contraceptive method compared to women receiving routine care.

The study population consists of pregnant women seeking a first trimester suction procedure in a single Medicaid-based practice in New York City. We need 125 participants in both the control group and the intervention group for a total of 250 participants. The inclusion criteria for enrollment in the study are (1) age greater than or equal to 18 years,(2) seeking contraception, (3) Spanish or English speaking, (4) access to a telephone, and (5) willing to participate in the study. We recognize that patients may be anxious about their scheduled procedure. Information about the procedure will be available to all patients in our clinic to inform and help alleviate anxiety.

After being consented, all participants will complete the baseline questionnaire. Participants will then be randomized in a 1:1 ratio.

Those randomized to the control group will proceed to routine care. Routine care consists of contraceptive counseling by the clinician performing the vacuum procedure. The clinician will evaluate the medical eligibility of each participant for FDA-approved contraceptive methods as part of routine care. Every clinician in the practice is a faculty member, fellow, or resident physician training under faculty supervision.

Those randomized to the intervention group will engage in structured counseling with the research coordinator, and then proceed to routine care. The structured counseling will take place while the participant would normally be waiting for care. We will pay attention to ensure that study participation does not prolong the clinic visit.

Structured counseling consists of a bilingual research coordinator going through the 2005 Decision Making Tool (D.M.T.) for family planning clients and providers developed by the World Health Organization(W.H.O.). Samples of each FDA-approved method will be present during the structured counseling session for participants to directly see and touch as desired. The link to this freely available counseling tool in English and Spanish is www.who.int/reproductivehealth/publications/dmt/index.html.

For our study, we modified the original version to include only FDA-approved contraceptive methods available in the United States suitable for a post-abortion population. Information about methods not available in the United States(NETEN injections, monthly injections and norplant) was removed. Information about new FDA-approved methods available in the United States (contraceptive patch, contraceptive ring, levonorgestrel IUS, and etonogestrel implant),but not previously included, was added. Information about methods not appropriate for post abortion patients (lactational amenorrhea and fertility awareness) was removed. We performed all modifications with the full support and cooperation of Sarah Johnson, technical officer in the Department of Reproductive Health and Research at the World Health Organization. We have attached our modified version with this application.

All FDA-approved methods will be available to participants on the day of their scheduled procedure for immediate initiation. Participants choosing an intrauterine device or implant will be able to have them placed that day.

Participants choosing depot medroxyprogesterone acetate will be able to have the injection that day. Participants choosing the pill, ring, or patch will receive a one month supply and continuing prescription that day. All participants will receive condoms and information about emergency contraception.

At the end of the visit, we will perform a brief secondary questionnaire. We will ask participants to indicate their chosen FDA-approved method and identify if the method was initiated that day.

Follow-up will take place at three months and six months with phone calls to obtain data from participants about the contraceptive method adopted and the contraceptive method use since enrollment.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* seeking contraception
* Spanish or English speaking
* has access to a telephone
* willing to participate in the study

Exclusion Criteria:

* age less than 18 years
* not fluent in English or Spanish
* not able to have access to a phone
* not seeking contraception

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2008-10; Primary Completion 2009-07 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Choice of contraceptive method on day of enrollment. | Day of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Westhoff, MD, MSc, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States